CLINICAL TRIAL: NCT06256679
Title: SUPERIOR HYPOGASTRIC PLEXUS PULSED RADIOFREQUENCY COMBINED WITH POSTERIOR TIBIALIS NERVE TRANSCUTANEOUS RADIOFREQUENCY AS A TREATMENT OPTION OF CHRONIC PELVIC PAIN MANAGEMENT IN INTERSTITIAL CYSTITIS
Brief Title: RADIOFREQUENCY TREATMENT OF CHRONIC PELVIC PAIN MANAGEMENT IN INTERSTITIAL CYSTITIS
Status: Completed | Type: Observational
Sponsor: Turkish League Against Rheumatism (Other)
Responsible Party: Principal Investigator, Muhammet Uğur ÖZTÜRK, Medical Doctor, Turkish League Against Rheumatism
Other Study IDs: TRASD- SUPERIOR HYPOGASTRIC
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Interstitial Cystitis, Chronic
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: SHP pulsed radiofrequency and TTNS: Patients with interstitial cystitis who received superior hypogastric plexus pulsed radiofrequency and transcutaneous tibial nerve stimulation.
  Interventions: Procedure: superior hypogastric plexus pulsed radiofrequency and transcutaneous tibial nerve stimulation
- Group 2: SHP pulsed radiofrequency: Group 2 included patients with interstitial cystitis who received only superior hypogastric plexus pulsed radiofrequency.
  Interventions: Procedure: superior hypogastric plexus pulsed radiofrequency

INTERVENTIONS:
Procedure: superior hypogastric plexus pulsed radiofrequency and transcutaneous tibial nerve stimulation — The L5-S1 intervertebral space was visualized using fluoroscopy. A 22G, 15 cm injection needle was advanced along the bilateral disc, and under lateral imaging, the needle position was confirmed anterior to the vertebral bodies. 2 ml of contrast solution was injected to confirm the correct needle placement, and then 8 mg of dexamethasone and 40 mg of bupivacaine (0.25%) were injected separately on each side. Two weeks later, patients who showed more than 50% improvement from the diagnostic block, as assessed by NRS, underwent a superior hypogastric pulsed radiofrequency procedure using a transdiscal technique with a 22G, 15 cm, 10 mm active-tipped radiofrequency needle at 42°C for 120 seconds. Two 50x50 mm electrode pads were placed on the posterior-superior aspect of the medial malleolus for posterior tibial nerve stimulation. Stimulation was delivered in continuous mode at a frequency of 20 Hz and a pulsed width of 200 ms. It was applied once a week for 30 min for 4 weeks.
  Groups: Group 1: SHP pulsed radiofrequency and TTNS
Procedure: superior hypogastric plexus pulsed radiofrequency — The L5-S1 intervertebral space was visualized using fluoroscopy. A 22G, 15 cm injection needle was advanced along the bilateral disc, and under lateral imaging, the needle position was confirmed anterior to the vertebral bodies.
  After negative aspiration of blood, 2 ml of contrast solution was injected to confirm the correct needle placement, and then 8 mg of dexamethasone and 40 mg of bupivacaine (0.25%) were injected separately on each side.
  Two weeks later, patients who showed more than 50% improvement from the diagnostic block, as assessed by NRS, underwent a superior hypogastric pulsed radiofrequency procedure using a trans discal technique with a 22G, 15 cm, 10 mm active-tipped radiofrequency needle at 42°C for 120 seconds.
  Groups: Group 2: SHP pulsed radiofrequency

SUMMARY:
Interstitial cystitis/painful bladder syndrome is a collection of symptoms that includes urinary urgency, urge incontinence, nocturia, and painful urination. Various treatment modalities are utilized in the management of the disease. Superior hypogastric plexus block, which is used in the treatment of chronic pelvic pain, is one of these treatment methods. Additionally, tibial nerve stimulation is used in the treatment of urinary symptoms. This study aims to compare the effectiveness of superior hypogastric plexus pulsed radiofrequency and adjunctive transcutaneous tibial nerve stimulation in the treatment of patients with interstitial cystitis

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Diagnosed with interstitial cystitis and experiencing symptoms for at least 3 months

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients with renal, hepatic, cardiovascular, or psychiatric diseases
* Additional interventional treatments within the first 3 months after the procedure
* A history of previous surgery or trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 34 patients diagnosed with interstitial cystitis by the urology department and experiencing symptoms for at least 3 months, who had undergone superior hypogastric nerve pulsed radiofrequency by our team, were retrospectively included in the study at the Algology Clinic of Hacettepe University Faculty of Medicine. Some of these patients had also undergone transcutaneous posterior tibial nerve stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Pre-intervention, 1st month, 3rd month
  NRS is a scale used to evaluate pain severity. Pain severity is evaluated between 0 and 10. A high score indicates a bad result.
Neuropathic Pain 4 Questions (DN4) | Pre-intervention, 1st month, 3rd month
  DN4 is a screening questionnaire to help identify neuropathic pain in clinical practice and research.
  This leads to a score range of 0-10 when the symptoms (range 0-7 points) as well as the signs (range 0-3 points) items are included. A high score indicates a bad result.
The O'Leary-Sant Interstitial Cystitis Symptom Index (ICSI) | Pre-intervention, 1st month, 3rd month
  The ICSI contains 4 items that measure urgency and frequency of urination, nighttime urination, and pain or burning. The ICSI score is is evaluated between 0 and 20. A high score indicates a bad result.
Interstitial Cystitis Problem Index (ICPI) | Pre-intervention, 1st month, 3rd month
  ICPI is a form that investigates how much problems the symptoms of interstitial cystitis cause. ICPI score is evaluated between 0 and 16. A high score indicates a bad result.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Medicine, Ankara, Turkey (Türkiye)